CLINICAL TRIAL: NCT00806689
Title: Full Disclosure Observational Cardiac Rhythm Documentation Follow-up After Surgical Atrial Fibrillation Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Luebeck (Other)
Responsible Party: Prof. Dr. med. Hans-H. Sievers, Clinic for Cardiac and Thoracic Vascular Surgery, University of Luebeck
Other Study IDs: 08-046
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2008-12

CONDITIONS: Atrial Fibrillation
Keywords: heart rhythm surveillance; follow-up; atrial fibrillation success
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery patients: Patients in atrial fibrillation being scheduled for cardiac surgery and concomitant ablation procedure
  Interventions: Procedure: Cardiac rhythm monitor implantation; Device: Reveal® XT 9525

INTERVENTIONS:
Procedure: Cardiac rhythm monitor implantation — post surgical procedure implantation of insertable event recorder for long time heart rhythm surveillance afte ablation therapy
  Other Names: Reveal® XT 9525, Medtronic Inc., Minneapolis, MN, USA
Device: Reveal® XT 9525 — During cardiac surgery after stand alone or concomitant ablation procedure, an insertable loop recorder will be implanted subcutaneously in left pectoral region. After surgery, patients will be monitored regularly in a quarterly basis by performing telemetry of the device in the outpatient clinic. Furthermore, home telemetry will be performed once a month for optimal heart rhythm observation.

SUMMARY:
24 hour Holter monitoring (24HM) is commonly used to assess cardiac rhythm after surgical therapy of atrial fibrillation. This "snapshot" rhythm documentation leaves a large diagnostic window of non recorded atrial arrhythmias and as such a large amount of uncertainty in follow-up result assessment. To improve accuracy of rhythm surveillance thus gaining a more "real-life" scenario of post surgical ablation therapy cardiac rhythm a new insertable cardiac rhythm monitor device (Reveal® XT 9525, Medtronic Inc., Minneapolis, MN, USA) with full observational continuous heart rhythm documentation is implanted.

In order to verify different follow-up strategies after surgical atrial fibrillation therapy, a comparison of different follow-up scenarios (symptoms, different cardiac documentation devices i.e. ECG and 24 hour Holter monitor, at different follow-up time points) is performed intraindividually. Thus the reliability of these devices and follow-up strategies to define success after ablation therapy is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients in atrial fibrillation (AF duration >4 months)being scheduled for cardiac surgery
* patients with lone atrial fibrillation being scheduled for surgical AF treatment

Exclusion Criteria:

* failure to provide informed consent
* current participation in another clinical trial
* organic cause of atrial fibrillation (hyperthyroidism etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who are scheduled for cardiac surgery and who also present with any kind of atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-12 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden development after surgical ablation therapy | 3 years

SECONDARY OUTCOMES:
Comparison of different cardiac rhythm documentation strategies to define success after ablation therapy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans-H. Sievers, M.D., Study Director — Clinic for Cardiac and Thoracic Vascular Surgery, University of Luebeck, germany; Thorsten Hanke, M.D., Principal Investigator — Clinic for Cardiac and Thoracic Vascular Surgery, University of Luebeck, germany; Ulrich Stierle, M.D., Study Chair — Clinic for Cardiac and Thoracic Vascular Surgery, University of Luebeck, Germany
Locations (1):
- Clinic for Cardiac and Thoracic Vascular Surgery, University of Lübeck, Germany, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Result] Hanke T, Charitos EI, Stierle U, Karluss A, Kraatz E, Graf B, Hagemann A, Misfeld M, Sievers HH. Twenty-four-hour holter monitor follow-up does not provide accurate heart rhythm status after surgical atrial fibrillation ablation therapy: up to 12 months experience with a novel permanently implantable heart rhythm monitor device. Circulation. 2009 Sep 15;120(11 Suppl):S177-84. doi: 10.1161/CIRCULATIONAHA.108.838474. PMID 19752365
- [Derived] Charitos EI, Ziegler PD, Stierle U, Robinson DR, Graf B, Sievers HH, Hanke T. Atrial fibrillation burden estimates derived from intermittent rhythm monitoring are unreliable estimates of the true atrial fibrillation burden. Pacing Clin Electrophysiol. 2014 Sep;37(9):1210-8. doi: 10.1111/pace.12389. Epub 2014 Mar 25. PMID 24665972
- [Derived] Charitos EI, Ziegler PD, Stierle U, Robinson DR, Graf B, Sievers HH, Hanke T. How often should we monitor for reliable detection of atrial fibrillation recurrence? Efficiency considerations and implications for study design. PLoS One. 2014 Feb 12;9(2):e89022. doi: 10.1371/journal.pone.0089022. eCollection 2014. PMID 24563690
- [Derived] Charitos EI, Stierle U, Ziegler PD, Baldewig M, Robinson DR, Sievers HH, Hanke T. A comprehensive evaluation of rhythm monitoring strategies for the detection of atrial fibrillation recurrence: insights from 647 continuously monitored patients and implications for monitoring after therapeutic interventions. Circulation. 2012 Aug 14;126(7):806-14. doi: 10.1161/CIRCULATIONAHA.112.098079. Epub 2012 Jul 23. PMID 22824434